CLINICAL TRIAL: NCT01687699
Title: Effects of Spironolactone on Cardio- and Cerebrovascular Morbidity and Mortality in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dialysis Outcomes Heart Failure Aldactone Study Group (Other)
Responsible Party: Principal Investigator, Yoshihiro Matsumoto, MD., PhD., Dialysis Outcomes Heart Failure Aldactone Study Group
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: dohas01
Record Dates: First submitted 2012-09-12; First posted 2012-09-19 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: End-stage Renal Failure
Keywords: cardiovascular event; hemodialysis; spironolactone
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- spironolactone (Experimental)
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: Spironolactone

SUMMARY:
Aldosterone receptor blockers reduce cardiac-related morbidity and mortality. Recently, we demonstrated that long-term low-dose spironolactone is clinically safe in many hemodialysis (HD) patients. In the present study, we assess whether low-dose spironolactone treatment reduces the high incidence of cardio- and cerebrovascular (CCV) morbidity and mortality in HD patients. The investigators' hypothesis is that aldosterone receptor blockade by spironolactone reduces the risk of both CCV morbidity and death among HD patients.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patients undergoing 4-hour-long HD thrice a week for at least 2 years
* With an average serum potassium level (immediately before dialysis on the first day of the week) of <6.5 mEq/l over the previous 2 months
* With a 24-hour urine output of <500 ml

Exclusion Criteria:

* A history of noncompliance
* Unstable vascular access
* Hypotension
* Hepatic failure
* Active cancer
* Any life-threatening disease other than ESRD

Min Age: 30 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
cardio- and cerebrovascular events

SECONDARY OUTCOMES:
death from all causes

CONTACTS AND LOCATIONS:
Locations (1):
- Shibukawa Clinic, Shizuoka, Shizuoka, Japan

REFERENCES:
- [Derived] Hasegawa T, Nishiwaki H, Ota E, Levack WM, Noma H. Aldosterone antagonists for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2021 Feb 15;2(2):CD013109. doi: 10.1002/14651858.CD013109.pub2. PMID 33586138
- [Derived] Matsumoto Y, Mori Y, Kageyama S, Arihara K, Sugiyama T, Ohmura H, Yakushigawa T, Sugiyama H, Shimada Y, Nojima Y, Shio N. Spironolactone reduces cardiovascular and cerebrovascular morbidity and mortality in hemodialysis patients. J Am Coll Cardiol. 2014 Feb 18;63(6):528-36. doi: 10.1016/j.jacc.2013.09.056. Epub 2013 Oct 30. PMID 24184249
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/19342857